CLINICAL TRIAL: NCT06689280
Title: Physical Rehabilitation of Older Persons Following a Community-Acquired Infection Hospitalization: A Feasibility Study
Brief Title: Physical Rehabilitation of Older Persons Following a Community-Acquired Infection Hospitalization - A Randomised-Controlled Trial
Acronym: REHAB-CAI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Birgitte Lindegaard Madsen, Associate professor, research responsible chief physician, PhD, Nordsjaellands Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REHAB-CAI (H-24047753)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Community-acquired Pneumonia; Urinary Tract Infections
Keywords: CAP; UTI
MeSH Terms: conditions — Community-Acquired Pneumonia; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-supervised home-based exercise training (Experimental): In-hospital exercise training: 30 min of daily one-on-one supervised exercise training using exercises from the exercise booklet "Sick but Healthy and Active".
  Patient-centred video-supervised home-based exercise intervention phase (weeks 0-12): 3 weekly exercise sessions (3 supervised sessions/week) over 12 weeks. Each session will last 45-50 min, consisting of 10-15 min of endurance, 20-30 min of resistance, and 5 min of balance exercises. The exercise intensity will progressively increase during the 12 weeks and be based on a target training intensity of 4-7 points on the Borg CR-10 scale. The exercise training is supplemented with weekly, individualised step-count goals that progressively increase (+5%) if previous step goals are achieved.
  Self-directed maintenance exercise phase (weeks 13-24): unsupervised self-directed exercise training 3 times per week for 12 weeks with phone calls, but with less frequency (see standard care below).
  Interventions: Behavioral: Video-supervised home-based exercise training
- Standard care (No Intervention): In-hospital: Patients will receive standard of care as recommended by their healthcare personnel.
  Control phase (weeks 0-12): Patients are contacted biweekly by phone calls after discharge up to 12 weeks after discharge. The patients will not receive any specific recommendations regarding physical activity.
  Control phase (week 13-24): The patients will continuously receive phone calls, but with less frequency (i.e., 3 calls per week in week 13-16, 1 call per week in week 17-20, and 0 call per week in week 21-24).

INTERVENTIONS:
Behavioral: Video-supervised home-based exercise training — 12 weeks of patient-centered video-supervised home-based exercise training that will be kick-started during hospitalization and continued for 12 weeks after discharge, followed by 12 weeks of self-directed maintenance exercise.
  Arms: Video-supervised home-based exercise training

SUMMARY:
Community-acquired infections such as community-acquired pneumonia (CAP) and urinary tract infection (UTI) remain leading causes of hospitalization and death due to infections in older persons in Europe. Hospitalization often results in further disabilities and frailty for older and frail individuals, from which some may never recover. Physical activity is well-established as a cornerstone in the primary prevention and treatment of several noncommunicable diseases. However, there is currently no established rehabilitation model following a pneumonia or other infection, nor is there any evidence to support the impact of rehabilitation on the mental and physical health of older and frail individuals following a pneumonia hospitalization or other infection.

The aim of the feasibility study is to evaluate a patient-centered and individualized exercise intervention that is kick-started during hospitalization and continued for 3 months after discharge with video-supervised home-based exercise training to patients hospitalized with CAP or UTI compared to standard care with regard to safety, clinical outcomes, patients' perception, functional ability, organizational aspects, and economic aspects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 years or 18-64 years if the presence of at least one chronic disease (e.g., diabetes, COPD, heart failure, etc.)
* Suspicious of a lower respiratory tract infection AND
* Presence of one or more symptoms of a lower respiratory tract infection such as fever ≥38.3°C, hypothermia <35.0°C, new onset of cough, pleuritic chest pain, dyspnea, or altered breath sounds on auscultation.
* Positive urine nitrate test and/or leukocyturia as depicted by positive esterase test or microscopy AND
* Presence of one or more symptoms of urinary tract infection such as dysuria, urgent or frequent urination, perineal or suprapubic pain, costo-vertebral tenderness or flank pain, fever (ear or rectal temperature of ≥38.2°C or axillary temperature of ≥38.0°C), or history of feeling feverish with shivering or rigors in the past 24 hours.
* Functionally independent before hospitalization and expected to be discharged to their own homes.
* Signed informed consent.

Exclusion Criteria:

* Hospitalization within the past 14 days.
* Inability to participate in the study due to dementia, paralysis, or other disorders.
* Severe aortic valve stenosis or terminal illness.
* Unstable cardiac arrhythmic disease.
* High risk for non-adherence as determined by screening evaluation.
* Already participating in regular exercise training.
* Unable to understand Danish.
* Unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-hospitalization (infection-related and all-cause) | 90 days after discharge.
  Report of the total number of re-hospitalized patients, defined as a hospital stay >12 hours.

SECONDARY OUTCOMES:
Re-hospitalization (infection-related and all-cause) | 30 days after discharge; 180 days after discharge.
  Report of the total number of re-hospitalized patients, defined as a hospital stay >12 hours.
Mortality (infection-related and all-cause) | 30 days after discharge; 90 days after discharge; 180 days after discharge; 360 days after discharge
  Report of the total number.
Handgrip strength | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Measure handgrip muscle strength in kilos in the dominant hand using a hand-held dynamometer. The highest number out of three attempts will be recorded.
Lower limb muscle strength and power | Baseline; 1-month after discharge (secondary endpoint), 3-month after discharge (primary endpoint), and 6-month after discharge (secondary endpoint).
  Assessment of muscle strength and power of the knee extensor muscles with dynamometry.
30-second sit to stand | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  A clinical test where the patient performs as many sit-to-stand actions as possible in 30 seconds. Measures leg muscle strength by counting the number of repetitions.
1-minute sit to stand | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  A clinical test where the patient performs as many sit-to-stand actions as possible in 1 minute. Measures endurance by counting the number of repetitions.
6-minute walking test | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Measure the distance in meters a person can walk in 6 minutes.
Short Physical Performance Battery (SPPB) | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  An objective measurement instrument combining 3 tests in 1 score. The tests consist of a balance test (measured in seconds), lower extremity strength (measured in seconds), and a walking test measuring functional capacity (measured in seconds).
Barthel index | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Measure of a persons ability to perform activities of daily living. Scores from 0 to 100. The higher the better.
Clinically Frailty Scale | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  A global clinical measure of the overall frailty of an older person. Scores from 1 to 9. The lower the better.
EuroQol-5D-5L (EQ-5D-5L) | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Measure health-related quality of life divided into the EQ-5D utility index and EQ-VAS score. The Danish EQ-5D-5L utility scores range from -0.757 for state 55555 to 1.0 for state 11111; the higher the score, the better. The EQ VAS is on a 0-100 scale; the higher the score, the better.
36-Item Short Form Survey (SF-36) | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Measure health-related quality of life. Total score from 0 to 100; the higher the score, the better.
COPD Assessment Test (CAT) | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  A patient self-administered questionnaire. An 8-item questionnaire designed to assess the impact of disease on a person's life (health status). Range of CAT scores from 0-40. Higher scores implicates a more severe impact of COPD on a patient's life (total score point).
Montreal Cognitive Assessment (MoCA) | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Measure of mild cognitive impairment. MoCa scores range from 0 to 30. Scores of 26 or over are considered to be normal.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); 6-month after discharge (secondary endpoint)
  A self-report rating scale that is designed to measure current symptoms of depression. Lower score is better.
Family Reported Outcome Measure (FROM-16) | 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); 6-month after discharge (secondary endpoint)
  Measure of the impact on the quality of life of an adult family member or partner resulting from having a person (of any age) in a family with any disease or condition, across all of medicine.
Physical activity level | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); 6-month after discharge (secondary endpoint)
  The objectivly measured physical activity level assessed with activity trackers.
Blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Concentration of p-phosphate (mmol/l), p-sodium (mmol/l), p-carbamide (mmol/l), and p-potassium (mmol/l).
Blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Concentration of pro- and anti-inflammatory cytokines (IL-6, Il-1ra, IL-18, IL-10, TNF-alpha, etc.)
Blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Concentration of lipids
Blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Concentration of galectin-3 (ng/ml), sST2 (ng/ml), and troponins (ng/ml).
Blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Concentration of NT-proBNP (ng/l).
Immune function | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Complete blood count with differential count. Concentration of immunoglobulin G (IgG), immunoglobulin M (IgM), and immunoglobulin A (IgA), and concentration of subclasses of IgG: IgG1, IgG2, IgG3, and IgG4.
Blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Concentration of HbA1c.
Blood sample | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); 6-month after discharge (secondary endpoint); and 12-month after discharge (secondary endpoint).
  Concentration of c-peptide (pmol/L).
Blood sample | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); 6-month after discharge (secondary endpoint); and 12-month after discharge (secondary endpoint).
  Concentration p-glucose (mmol/L).
Blood sample | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); 6-month after discharge (secondary endpoint); and 12-month after discharge (secondary endpoint).
  Concentration of p-insulin (pmol/L).
Biobank blood sample | Baseline; discharge (secondary endpoint); 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), 6-month after discharge (secondary endpoint), and 12-month after discharge (secondary endpoint).
  Whole blood, plasma, and serum.
Insulin resistance | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint), and 6-month after discharge (secondary endpoint).
  The Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) will be used to measure severity of insulin resistance. Normal reference levels for HOMA-IR is 0.7 to 2.0, with values >2.0 representing clinically significant insulin resistance.
Glycemic variability | Baseline (day 0-10); 3-month after discharge (day 80-90, primary endpoint), and 6-month after discharge (day 170-180, secondary endpoint).
  Glucose outcomes from the CGM sensor (Dexcom G6) including time in range (TIR) for blood glucose, time above range (TAR) for blood glucose, time below range (TBR) for blood glucose, average blood glucose, and variance in blood glucose (CV).
P-glucose during an oral glucose tolerance test (OGTT) | Baseline; 3-month after discharge (primary endpoint), and 6-month after discharge (secondary endpoint).
  P-glucose (mmol/L) measured during an OGTT.
P-insulin during an oral glucose tolerance test (OGTT) | Baseline; 3-month after discharge (primary endpoint), and 6-month after discharge (secondary endpoint).
  P-insulin (pmol/L) measured during an OGTT.
C-peptide during an oral glucose tolerance test (OGTT) | Baseline; 3-month after discharge (primary endpoint), and 6-month after discharge (secondary endpoint).
  C-peptide (pmol/L) measured during an OGTT.
Insulin sensitivity | Baseline; 3 month after discharge (primary endpoint); 6 months after discharge (secondary endpoint).
  Insulin sensitivity using Matsuda index. The index is calculated based on p-glucose and p-insulin in fasting state and during an OGTT.
Glucose-lowering medication | Baseline; 3 months after discharge (primary endpoint); 6 months after discharge (secondary endpoint)
  Changes in glucose-lowering medication in patients with diabetes
Semi-structured qualitative interviews | 1-month after discharge (seconary endpoint), 3-month after discharge (primary endpoint), and 6-month after discharge (secondary endpoint).
  Semi-structured qualitative interviews with the patient and a relative. The following themes will be explored: perception of the content in the exercise intervention, barriers and enablers towards physical activity, ideas for improvement of the exercise intervention
Adverse events | At 1-month after discharge, 3-month after discharge (primary endpoint), and 6-month after discharge.
  Numbers of severe adverse events and adverse events
Total and appendicular lean and fat mass | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  DXA-scan
Muslce quality and density | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Midt-thigh CT-scan
Fat mass index and fat-free mass index | Baseline; 1-month after discharge (secondary endpoint); 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Bioelectrical impedance analysis
Muscle oxidative stress and inflammation | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Muscle biopsies from the m. vastus lateralis of the quadriceps muscle
Muscle protein synthesis and proteolysis | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Muscle biopsies from the m. vastus lateralis of the quadriceps muscle
Muscle insulin sensitivity | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint).
  Muscle biopsies from the m. vastus lateralis of the quadriceps muscle
Skeletal muscle cell growth, development, and function | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint)
  Skeletal muscle cell cultures of muscle tissue from m. vastus lateralis of the quadriceps muscle.
Insulin sensitivity and signaling of adipose tissue | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (secondary endpoint)
  Adipose tissue biopsy
Adipose tissue inflammation | Baseline; 3-month after discharge (primary endpoint); and 6-month after discharge (seconary endpoint)
  Adipose tissue biopsy
Adipose tissue immune cell infiltration | Baseline; 3-month after discharg (primary endpoint); and 6-month after discharge (secondary endpoint)
  Adipose tissue biopsy
Pulmonary medication | Baseline; 3 months after discharge (primary endpoint); 6 months after discharge (secondary endpoint)
  Changes in pulmonary medication (tablets and inhalation)
Lung function | Baseline; 3 months after discharge (primary endpoint); 6 months after discharge (secondary endpoint)
  Spirometry in patients with COPD
Lung function | Baseline; 3 months after discharge (primary endpoint); 6 months after discharge (secondary endpoint)
  Body plethysmography in patients with COPD
Lung function | Baseline, 3 months after discharge (primary endpoint); 6 months after discharge (seconary endpoint)
  Single-breath carbon monoxide uptake in patients with COPD
Acute exacerbations of COPD | Baseline; 3 months after discharge (primary endpoint); 6 months after discharge (secondary endpoint)
  Notification of acute exacerbations of COPD through patient files
Health economics | From baseline to 360 days after discharge.
  Health costs, the cost per quality-adjusted life years (QALYs), and the lifetime estimated cost per QALY gained will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Lindegaard, MD, PhD, Principal Investigator — Department of Pulmonary and Infectious Diseases, Copenhagen University Hospital - North Zealand
Locations (3):
- Denmark (3):
  - Department of Pulmonary and Infectious Diseases, Copenhagen University Hospital, Hillerød
  - Department of Infectious Diseases, Copenhagen University Hospital, Amager-Hvidovre, Hvidovre
  - Department of Respiratory Medicine, Copenhagen University Hospital, Amager-Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: No